CLINICAL TRIAL: NCT05057754
Title: Enhancing Sonographic Measurement of Intraneural Blood Flow in the Median Nerve
Brief Title: Sonographic Measurement of Intraneural Blood Flow in the Median Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Shawn Roll, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS-21-04511
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Carpal Tunnel Syndrome; Median Nerve Injury
Keywords: intraneural blood flow
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Cool-Down Exercise; Heating; Cooking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): A total of 50 participants are estimated to be recruited, each completing six conditions in the following order: 1) wrist cooling, 2) wrist heating, 3) exercising, 4) typing, 5) using a mouse, 6) cooking, with an observation of intraneural blood flow assessed with Doppler sonography before and after each condition.
  Interventions: Behavioral: Cooling; Behavioral: Heating; Behavioral: Exercising; Behavioral: Typing; Behavioral: Using a mouse; Behavioral: Cooking

INTERVENTIONS:
Behavioral: Cooling — Participants' dominant hand and wrist will be immersed in cool water (20°C) for five minutes. The cool water will be kept to around 20°C (19 - 21°C) by frequently checking the temperature and corrected when it rises to 20.5°C
Behavioral: Heating — A heat pack wrapped in a towel will be applied to participants' dominant hand for five minutes.
Behavioral: Exercising — Participants will be asked to participate in moderate-intensity physical activities to induce an increase in blood pressure. The physical activity will be two sets of 30 jumping jacks, followed by 15 squats. Participants are allowed to rest for 20 seconds between the two sets.
Behavioral: Typing — All participants will be asked to perform a typing task with a standard wired keyboard. All subjects will be asked to type for five minutes.
Behavioral: Using a mouse — Participants will be asked to draw as many lower-case alphabet characters from "a" to "z" as possible using a standardized scroll mouse for five minutes in the Windows Microsoft Paint software.
Behavioral: Cooking — Participants will be asked to participate in a cooking trial following a prespecified cooking recipe of Rice Krispy Treat. he participant will be asked to follow the procedures as follows: (1) cut and put wax paper in the pan; (2) cut butter into 4 pieces; (3) place butter in a pot over a portable stove and stir until the butter is completely melted; (4) add four oz of marshmallows and stir until melted; (5) add cereal and the rest of marshmallows and stir until all ingredients are combined (6) transfer the ingredients to the pan and use a silicone spatula to pat the ingredients evenly into pan.

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common nerve compression disease and the most expensive upper-extremity work-related musculoskeletal disorder, affecting approximately 10 million people in the US. To understand the clear etiology and mechanism of carpal tunnel syndrome, the measurement of median nerve intraneural blood flow needs to be further scrutinized as the common fluctuating physiological conditions and functional hand activities might contribute to the fluctuation of the measurement and serve as measurement error. This study aims to examine how intraneural blood flow within the median nerve is affected by physiological factors (i.e., body temperature and blood pressure) and functional hand activities (i.e., typing, using a mouse, and cooking).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65
* English-speaking
* Ability to endure a moderate-intensity physical activity
* Ability to type without looking at the keyboard

Exclusion Criteria:

* Pain, tingling, or numbness in the hand or wrist region within the past week
* History of corticoid injection in the upper extremity
* History of surgery in the wrist region
* Carpal tunnel syndrome
* Amyotrophic lateral sclerosis
* Diabetes
* Hypothyroidism
* Pregnant
* Positive Phalen's test
* Persistent median artery within wrist region
* Bifid median nerve

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Change in intraneural blood flow after intervention | Immediately prior to and after each intervention
  Doppler ultrasound images will be repeatedly collected to obtain the primary outcome measure for this study, intraneural blood flow. After identifying the course of the median nerve in the longitudinal plane (I.e., the sagittal plane), intraneural blood flow at the level of carpal tunnel measured as the peak systolic velocity of the identified blood flow signal will be observed and collected.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn C Roll, PhD, Study Director — University of Southern California
Locations (2):
- United States (2):
  - USC; Musculoskeletal Sonography & Occupational Performance Laboratory, Los Angeles, California
  - Ohio State University; School of Health and Rehabilitation Sciences, Columbus, Ohio